CLINICAL TRIAL: NCT05283161
Title: CBD/THC Solution as a Pharmacological Strategy for Patients With Fibromyalgia. Single-center, Double-blind, Randomized, Placebo-controlled Clinical Trial Protocol (FibroCann)
Brief Title: CBD (Cannabidiol)/THC (Tetrahydrocannabinol) Solution as a Pharmacological Strategy for Patients With Fibromyalgia (FibroCann)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: FG Brasil LTDA (Industry)
Collaborators: 3F Clinical Trials LTDA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 04200240
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Fibromyalgia
Keywords: rheumatic syndrome; Muscle pain; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Myalgia | interventions — Cannabidiol; Dronabinol

STUDY DESIGN:
Intervention Model Description: This single center clinical trial is a double-blinded, randomized, placebo-controlled and dose-response type, having a pre-randomization period (8 days prior to the beginning of the study), and a 120-day double-blind main period. Patients will be double-blind randomized in a 1 by 1 by 1 by 1 ratio to receive cannabidiol and tetrahydrocannabinol 1 by 1: (0.1 mg/ml) (10 research participants), cannabidiol and tetrahydrocannabinol 1 by 1 (1.0 mg/ml) (n=10), cannabidiol and tetrahydrocannabinol 1 by 1 (10 mg/ml) (10 research participants) and placebo (vehicle) (10 research participants). The administration will occur daily, once a day, during the night period, before going to bed and 30 minutes after the meal, during the next 120 days. The clinical study will have a baseline assessment (T0), one day before the start of the intervention with the solution. The tools will be reapplied after 15 (T1), 30 (T2), 60 (T3), 90 (T4) and 120 (T5) days of intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo will match the study drug in odor, taste, color and appearance to ensure proper masking. Eligible patients included in the pre-randomization period will be double-blind randomized in a 1:1:1:1 ratio between the experimental groups, by a biostatistician who is not involved in data collection nor analysis, to receive the CBD/THC solution at doses of 0.1mg/day, 1mg/day, 10mg/day, or placebo. A randomization sequence will be generated by computer, which creates identification codes necessary for the correct labeling of the drug and allocation of the patients in the experimental groups (https://www.sealedenvelope.com). This code will be adopted in the Case Report Form of the patient. The designation of the experimental group will be known by the data analysts, but hidden from the participants and the team involved with the treatment and research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): 10 participants will receive placebo (vehicle). The placebo will match the study drug in odor, taste, color and appearance. The administration will occur daily, once a day, during the night period, before going to bed and 30 minutes after the meal, during the next 120 days.
  Interventions: Drug: Placebo
- cannabidiol and tetrahydrocannabinol 1:1 (0.1 mg/ml) (Experimental): 10 participants will receive CBD and THC in the same concentration (1:1) (0.1 mg/ml). The administration will occur daily, once a day, during the night period, before going to bed and 30 minutes after the meal, during the next 120 days.
  Interventions: Drug: cannabidiol and tetrahydrocannabinol
- cannabidiol and tetrahydrocannabinol 1:1 (1.0 mg/ml) (Experimental): 10 participants will receive CBD and THC in the same concentration (1:1) (1.0 mg/ml). The administration will occur daily, once a day, during the night period, before going to bed and 30 minutes after the meal, during the next 120 days.
  Interventions: Drug: cannabidiol and tetrahydrocannabinol
- cannabidiol and tetrahydrocannabinol 1:1 (10.0 mg/ml) (Experimental): 10 participants will receive CBD and THC in the same concentration (1:1) (10.0 mg/ml). The administration will occur daily, once a day, during the night period, before going to bed and 30 minutes after the meal, during the next 120 days.
  Interventions: Drug: cannabidiol and tetrahydrocannabinol

INTERVENTIONS:
Drug: cannabidiol and tetrahydrocannabinol — CBD and THC will be given in the same concentration within a group of 10 participants, while its effects will be compared with the other two groups with 10 participants each and the placebo group.
  Other Names: CBD/THC; CBD and THC
  Arms: cannabidiol and tetrahydrocannabinol 1:1 (0.1 mg/ml); cannabidiol and tetrahydrocannabinol 1:1 (1.0 mg/ml); cannabidiol and tetrahydrocannabinol 1:1 (10.0 mg/ml)
Drug: Placebo — The placebo will match the study drug in odor, taste, color and appearance to ensure proper masking.
  Arms: Placebo

SUMMARY:
Fibromyalgia is considered a chronic pain syndrome, non-inflammatory, of unknown etiology, which manifests itself in the musculoskeletal system in up to 2.5% of the general population, predominantly in females, mainly between 35 and 44 years old, having a direct impact on the quality of life of their patients (JUNIOR; GOLDENFUM; SIENA, 2012; HEYMANN et al., 2017). In 1990, eighteen (18) specific sites were defined as tender points which are used to better diagnose fibromyalgia (WOLFE et al., 2010). Due to its clinical and exclusion diagnosis, treatment usually starts late, which allows the progression of symptoms and corroborates its low efficiency in the long term (DE SOUSA BRAZ et al., 2011). Due to the ineffective results and significant side effects that conventional treatment with drugs such as antidepressants, analgesics and anti-inflammatory drugs can provide, patients, physicians and researchers are looking for new main or adjuvant treatments, pharmacological and non-pharmacological (DE SOUSA BRAZ et al. al., 2011). In this context, it has been seen that the use of Cannabis sativa as a therapeutic option in fibromyalgia is promising, especially in reducing the pain caused by the disease and also the adjuvant symptoms, such as depression and sleep disorders (YASSIN; ORON; ROBINSON, 2019). This result must occur due to the action of cannabinoids, such as CBD and THC, on cannabinoid receptors distributed in peripheral nerves, spinal cord and supraspinal region, sites responsible for the reception, transmission and perception of pain (STE-MARIE et al., 2012). Currently, cannabinoids are considered safe analgesics with considerable efficacy, which demonstrates potential as a therapeutic option in the treatment of chronic pain, particularly in patients refractory to other treatments (HAUSER et al., 2018). In addition to its action on the painful mechanisms of fibromyalgia, the antidepressant effects of Cannabis are of great value in the treatment of fibromyalgia. These effects are explained by the modulation on serotonin 5-HT1A receptors, which has its effect exerted especially by CBD (ESPEJO-PORRAS et al., 2013).

Considering that research has reported the effects of phytocannabinoids on the painful symptoms of fibromyalgia (HAUSER et al., 2018), the hypotheses of the present study are:

Primary hypothesis: The dose-response curve and ED50 for the primary outcome, which is related to pain intensity, will be determined in the dose range between 0.1 and 10mg/day. The sensation of pain will be significantly reduced in participants receiving oral solution containing CBD/THC 10mg/day compared to those who will receive placebo.

Secondary hypothesis: There will be a reduction in pain catastrophizing, as well as an improvement in the acceptance and action rate related to pain, a reduction in depression, an improvement in sleep latency and quality, a reduction in insomnia and an increase in the quality of life in patients treated with oral solution containing CBD/THC 10mg/day compared to those receiving placebo.

Supporting Hypothesis: The tested CBD/THC solution will show efficacy and safety with no serious adverse effects.

DETAILED DESCRIPTION:
Patients with fibromyalgia will be recruited from tertiary health care establishments, specifically patients treated in the area of rheumatology, for eligibility assessment according to inclusion and exclusion criteria by the rheumatologist participating in this study, Osvaldo Haider Jr (CRM- PR 22274). It is important to point out that the patients' participation in the study will be voluntary, with no expectation of remuneration of any kind.

Recruitment for the two stages will follow these steps:

The first recruitment, in tertiary health care centers, in the rheumatology specialty, will start after approval of this project by the ethics committee; Dissemination of the study will be carried out via social networks and direct dissemination to doctors and tertiary health care clinics, which serve the rheumatology specialty; Enrolled volunteers must attend the evaluation for the inclusion and exclusion criteria, which will be carried out at the 3F Clinical Trials research center in a reserved environment at the clinical research centers contracted by 3F Clinical Trials; Patients must come with a medical report attesting to the diagnosis of fibromyalgia; The clinical evaluation, to meet the inclusion and exclusion criteria, will be performed under the supervision of the Rheumatologist Principal Investigator (PI) of this study, Osvaldo Haider Jr (CRM-PR 22274). Assessments of clinical symptoms, history will be performed, and the patient will be referred for laboratory tests of renal and hepatic profile. Additionally, women of childbearing age will undergo a biochemical hCG test. Additional tests for diagnostic confirmation or confirmation of any inclusion and exclusion criteria from the study may be requested; If there is a need for analysis of exams or the patient's medical history, it will be formally requested to the tertiary care center, where the patient undergoes his regular treatment, according to the requirements of the place, and according to the data use term. on file, the data will be kept confidential; Patients who are able to participate in the study, according to a clinical rheumatological evaluation, will undergo a pharmaceutical evaluation, carried out by the pharmacist responsible for this study, Ma. Ana Carolina Martins (e-CRF-PR 29255), to analyze the criteria in relation to the previous use of Cannabis, drug interactions in conventional treatment, possible reports that may exclude the patient from the study; Being able to participate in the study, the selected patients must read the informed consent; Patients will be informed that the project is placebo-controlled, and that this allocation to active treatment or placebo is random and double-blind; Agreeing with the terms, the patient will sign the informed consent in two copies, one for him and another for the researcher.

Participants will undergo a variety of examinations, questionnaires and tests during screening, enrollment and allocation, in-intervention assessments, final treatment assessment and for a post-trial period monitoring period. It is noteworthy that the evaluations performed through the clinical questionnaires established in this protocol will be made by telephone.

The following tests and protocols will be used: Pregnancy Test and Vital Signs; Pain; Depression; Sleep; Quality of life; Adverse Effects Monitoring; Laboratory; Tests.

The pre-randomization period will take place in weeks -8 to 0 in order to make sure that all participants meet all the inclusion criteria. Participants who are under pharmacological treatment must have their treatments stable for at least 60 days and not make changes to these treatments during the clinical trial, without such procedure being duly registered.

Patients eligible for the study, following the inclusion and exclusion criteria, will be randomized in a 1:1:1:1 ratio to receive CBD/THC 1:1 (0.1 mg/ml) (n=10), CBD/THC 1:1 (1.0 mg/ml) (n=10), CBD/THC 1:1 (10 mg/ml) (n=10) or placebo (vehicle) (n=10), daily, once a day day. The treatment will have a total duration of 120 days.

The dose was chosen based on preliminary results of pilot studies conducted by this research group (with unpublished results) and also according to the characteristics of the drug produced by the sponsor. In addition, evidence has shown that doses in previously published studies have doses within this range or even above the concentration determined for our study (see item 11.1).

The clinical study will have a baseline assessment (T0), one day before the start of the intervention with the solution. The tools will be reapplied after 15 (T1), 30 (T2), 60 (T3), 90 (T4) and 120 (T5) days of intervention. Medical monitoring of vital signs and clinical evidence of potential adverse effects will take place throughout the study. In this trial, for ethical reasons, patients will not be advised to discontinue the pharmacological treatment currently in use (e.g., opioids, antidepressants, benzodiazepines, gabapentinoids, anti-inflammatory drugs, or other non-opioid analgesics).

The CBD/THC solution will be administered to participants as an oral solution. The drug will be provided by the company FG Brasil LTDA, under the trade name Aura Pharma, which is a company that imports cannabinoid products and sponsors this study.

The product consists of a solution containing the phytopharmaceuticals CBD and THC, both at a concentration of 10mg/mL. The dilution vehicle is MCT (medium chain triglycerides) oil. Product development is carried out at Schibano Pharma AG Tüfi, 450 - Wald Schönengrund - 9105, Switzerland, and is obtained under Good Manufacturing Practices (GMP) protocols, ensuring a level of pharmaceutical quality for human use, and free from the addition of isolated substances of synthetic or semi-synthetic origin.

The sponsor will also provide the placebo, which consists of the vehicle without the addition of CBD and THC phytopharmaceuticals, maintaining the same organoleptic aspects of the CBD/THC solution.

The solution will be provided by the study sponsor, packaged in 10 mL vials, along with a dosing syringe (with graduation lines) for oral administration. The patient will be instructed to store the bottle in a place with a temperature of up to 30°C, dry, protected from light and heat, and out of the reach of children.

Dilution will be carried out in the same vehicle as the base drug, which will be provided by the sponsor, for doses of 0.1 and 1mg/ml. Thus, all patients will aspirate the equivalent volume to be administered (1mL/day) from their own bottle, corresponding to: (i) Group 1: 0.1mg of CBD and 0.1mg of THC; (ii) Group 2: 1mg of CBD and 1mg of THC; (iii) Group 3: 10mg of CBD and 10mg of THC; (iv) Group 4: placebo/vehicle. The time of administration will be daily, in the evening before going to bed, and 30 minutes after the meal. Participants will be instructed to wash the syringe with water and detergent after use, and rinse thoroughly with running water through repetitive aspirations.

It should be noted that a double quality control will be carried out, with physical-chemical analysis, prior to the availability of the product for the study. The first quality review is carried out by the product developer in Switzerland. Finally, the second quality analysis is performed by Aura Pharma in Brazil.

Labeling and storage:

All study products will be labeled in English and Portuguese in accordance with local regulations for investigational drugs.

A total of 40 patients will be required to detect a significant difference from treatment with the standardized CBD/THC solution. We performed an a priori calculation using the effect size described by Yanes et al. (2019) (Cohen's d = 0.58), considering an analysis of covariance (ANCOVA) design for repeated measures, alpha (α) set at 5% and statistical power (β) at 80%. In this case, we use the software GPower* 3.1.9.7 (Heinrich-Heine-Universityät, Düsserldorf). The collection and preservation of clinical data complies with standard requirements for data management and handling in accordance with the ICH/BPC. A secure database will be established for the collection of clinical data through the e-CRF platform via a secure connection at clinical research facilities and with traceable restricted access. All data obtained during the study will be documented in the individual e-CRF. In case of missing data, the reasons for this will be noted in the e-CRF.

Participant information collected in the e-CRF, but not recorded in the patient's files, will be considered as source documents. Patient participation and any treatment-related AE in the study will be documented in the e-CRF. No patient information, such as medical history and medication history, will be collected before the informed consent has been obtained from the patient. Information obtained directly from potential participants prior to obtaining the informed consent (ie, during eligibility screening) will be recorded in the e-CFR, and this information will be made available to researchers with the patients' permission.

The study will end when the last patient completes the last clinical evaluation at the end of 120 days of treatment, or the patient may for some reason discontinue the intervention and choose to withdraw from the clinical trial. This protocol will be suspended or terminated if the Principal Investigator, in agreement with the research team: Perceive that there is a risk or harm to the health of voluntary participants, and this risk is directly associated with the investigational drug and not provided in the informed consent; observe the occurrence of a serious adverse event after signing the informed consent, which results in: 1) death; 2) threat or risk to life; 3) need for hospitalization; 4) prolongation of preexisting hospitalization; 5) permanent disability or damage; or 6) a significant medical occurrence that, based on appropriate medical judgment, may impair the participant's exclusion criteria and/or require medical or surgical intervention to prevent any of the other aforementioned occurrences. In case of termination or suspension of this study, all participants will be informed, receive appropriate therapy and be followed up by the responsible physician and research team.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of fibromyalgia based on the pharmacological criteria of the American College of Rheumatology, 2016 to fibromyalgia, having received three months of pharmacological treatment without relevant clinical improvement;
* Adult individuals (aged 18 to 75 years) with a mean pain intensity greater than or equal to 7 on the FIQ numerical pain scale (Fibromyalgia Impact Questionnaire);
* No use of Cannabis or its derivatives (THC and CBD) in any systemic administration route in the last six months;
* Capability to read, write and speak in Portuguese (Brazil);
* Sign the ICF (Informed Consent Form).

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Any known pathology, in an advanced stage, associated with the locomotor system (arthritis, osteoarthritis, uric acid);
* Neurological disorders;
* Previously reported renal disorders or changes in the exams during the pre-randomization stage;
* Previously reported liver disorders or changes in tests during the pre-randomization stage;
* Peripheral neuropathy;
* Known serious cardiovascular disease (uncontrolled hypertension, heart failure, cardiac pacemaker);
* Medical decision that participation in the study is not in the best interest of the patient;
* Making previous use of cannabinoids by any route of administration;
* Diagnosis of alcohol dependence;
* Usage of psychotomimetic drugs or narcotics;
* Having participated in research projects in the two months prior to the beginning of the study;
* Having a history or having first-degree relatives with a history of psychosis in any level at least once in their lifetime;
* Inappropriate metabolic profile of THC or CBD cannabinoids for the use of the test doses in this study, observed by pharmacogenetic testing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2022-08-20 (Estimated); Study Completion 2022-11-20 (Estimated)

PRIMARY OUTCOMES:
Dose-response curve and median effective dose | Within 120 days
  The primary outcome is the dose-response curve and median effective dose (ED50) in relation to the change in pain intensity within the dose range determined in this study, compared to placebo, as measured by the McGill Questionnaire.

SECONDARY OUTCOMES:
Pain catastrophizing | Within 120 days
  Effectiveness in changing fibromyalgia symptoms through a change in pain catastrophizing: by the Pain Catastrophic Scale (B-PCS). A questionnaire is applied to patients aiming to indicate the degree to which they have thoughts and feelings when they are experiencing pain using the 0 (not at all), 1 (to a slight degree), 2 (to a moderate degree), 3 (to a great degree) and 4 (all the time) scale. A total score is yielded (ranging from 0-52), along with three subscale scores assessing rumination, magnification and helplessness. A total PCS score of 30 represents clinically relevant level of catastrophizing.
Acceptance in relation to pain | Within 120 days
  Change of acceptance and daily action in relation to pain: by the Acceptance and Action Questionnaire-II (AAQ-II). A questionnaire containing statements is applied to patients aiming to indicate the degree to which they have thoughts and feelings when they are experiencing pain using the 1 (never true), 2 (very seldom true), 3 (seldom true), 4 (sometimes true), 5 (frequently true), 6 (almost always true), 7 (always true). The association of the score values with the acceptance to pain will vary with the statements in the questionnaire.
Depressive symptoms | Within 120 days
  Change in depressive symptoms: data from the Beck Depression Inventory and the Hamilton Depression Rating Scale (HAM-D). In both tests, higher scores are related to higher levels of depession. Generally, in the Beck Depression Inventory, scores 1-10 are considered normal; 11-16 are considered to be Mild mood disturbance; 17-20 are considered to be Borderline clinical depression; 21-30 are considered to be Moderate depression; 31-40 are considered to be Severe depression and values over 40 are considered as Extreme depression. In theHAM-D Scores: A pacient score around 0-7 is considered as Normal; 8-13 is considered as Mild; 14-18 is considered as Moderate; 19-22 is considered as Severe; ≥23 is considered as Very severe.
Sleep quality | Within 120 days
  Change in sleep quality: Subjective domain of sleep quality using the Pittsburgh Sleep Quality Index (PSQI). In the Pittsburgh Sleep Quality Index, nineteen individual items are used to generate seven considerations: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The scores for these seven components are summed to yield a total score ranging from 0 to 21, with the global score indicating worse sleep quality.
Insomnia Severity | Within 120 days
  By the Insomnia Severity Index; Change in quality of life: using the Fibromyalgia Impact Questionnaire (FIQ). The Insomnia Severity Index has seven questions. The scores for these seven components are summed to yield a total score. Results ranging from 0-7 mean no clinically significant insomnia; 8-14 mean subthreshold insomnia; 15-21 mean moderate severity insomnia; 22-28 mean severe insomnia. In the The Fibromyalgia Impact Questionnaire, higher score indicates a greater impact of the insomnia syndrome on the person.
Daytime sleepiness | Within 120 days
  Absence of daytime sleepiness: according to the Epworth sleepiness scale (ESS). The ESS is a self-administered questionnaire with 8 questions. The questions can be answered ranging 0 to 3, according to their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score is the sum of the values of the 8 questions and can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'. Generally scores ranging 0-5 mean Lower Normal Daytime Sleepiness; 6-10 mean Higher Normal Daytime Sleepiness; 11-12 mean Mild Excessive Daytime Sleepiness; 13-15 mean Moderate Excessive Daytime Sleepiness; 16-24 mean Severe Excessive Daytime Sleepiness.
Sleep duration | Within 120 days
  Change in sleep duration: PSQI, sleep duration domain

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Antonio H Junior, Principal Investigator — 3F Clinical Trials LTDA

IPD SHARING:
Plan to Share IPD: No